CLINICAL TRIAL: NCT02728102
Title: Phase II Multicenter Trial of Single Autologous Hematopoietic Cell Transplant Followed by Lenalidomide Maintenance for Multiple Myeloma With or Without Vaccination With Dendritic Cell/Myeloma Fusions (BMT CTN 1401)
Brief Title: Dendritic Cell/Myeloma Fusion Vaccine for Multiple Myeloma (BMT CTN 1401)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1401; U01HL069294 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Lenalidomide; Maintenance Therapy; Hematologic Disorders; Vaccine; GM-CSF; Transplant; Anti-Myeloma Agents
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases | interventions — Melphalan; Leukapheresis; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lenalidomide, vaccine, and GM-CSF (Experimental): Patients will undergo tumor cell collection and autologous stem cell transplant with melphalan. Patients will undergo leukapheresis and then will receive maintenance lenalidomide with myeloma vaccine and GM-CSF.
  Interventions: Procedure: Tumor Cell Collection; Procedure: Autologous Stem Cell Transplant; Drug: Melphalan; Procedure: Leukapheresis; Biological: Myeloma vaccine; Drug: GM-CSF; Drug: Lenalidomide
- Lenalidomide and GM-CSF (Active Comparator): Patients will undergo tumor cell collection and autologous stem cell transplant with melphalan. Patients will receive maintenance lenalidomide with GM-CSF.
  Interventions: Procedure: Tumor Cell Collection; Procedure: Autologous Stem Cell Transplant; Drug: Melphalan; Drug: GM-CSF; Drug: Lenalidomide
- Maintenance Lenalidomide (Active Comparator): Patients will undergo tumor cell collection and autologous stem cell transplant with melphalan. Patients will receive maintenance lenalidomide.
  Interventions: Procedure: Tumor Cell Collection; Procedure: Autologous Stem Cell Transplant; Drug: Melphalan; Drug: Lenalidomide

INTERVENTIONS:
Procedure: Tumor Cell Collection — Patients will undergo aspiration of 30 mL of bone marrow from which myeloma cell preparations will be generated. Myeloma cells will be isolated and frozen for subsequent vaccine generation for patients randomized to the vaccine arm (randomization occurs after transplant and recovery).
Procedure: Autologous Stem Cell Transplant — Patients will receive an autologous graft with a minimum cell dose of 2.0 x 10^6 CD34+ cells/kg patient actual body weight per autologous transplantation.
Drug: Melphalan — Autologous hematopoietic cell transplant will be done with high-dose melphalan of 200mg/m^2 at the schedule and timing according to institutional practices.
  Other Names: Alkeran
Procedure: Leukapheresis — Blood samples will be collected through a catheter in the neck or chest and leukapheresis will be performed using standard clinical procedures.
  Arms: Lenalidomide, vaccine, and GM-CSF
Biological: Myeloma vaccine — The target dose is 3 x 10^6 fusion cells per vaccine. A minimum of 3 x 10^6 total fusion cells will be required to proceed with vaccine administration. Patients who have <3 x 10^6 total fusion cells will not proceed with vaccination. Patients will receive the DC/MM fusion vaccine on day 1 of cycles 2, 3, and 4 of lenalidomide maintenance. Vaccine will be administered by subcutaneous injection in the upper thigh.
  Other Names: Dendritic cell fusion vaccine; DC/MM fusion vaccine
  Arms: Lenalidomide, vaccine, and GM-CSF
Drug: GM-CSF — 100 ug GM-CSF will be given subcutaneously in the upper thigh and daily for a total of 4 days of each cycle.
  Other Names: Granulocyte macrophage colony-stimulating factor; Leukine
  Arms: Lenalidomide and GM-CSF; Lenalidomide, vaccine, and GM-CSF
Drug: Lenalidomide — Maintenance therapy with lenalidomide will begin between 90 and 100 days after stem cell infusion. Lenalidomide will be administered initially at a dose of 10 mg per day continuously. Cycle duration during maintenance therapy is 28 days. Patients will continue lenalidomide for two years from initiation of therapy.
  Other Names: Revlimid™

SUMMARY:
The study is designed as a Phase II, multicenter trial of vaccination with Dendritic cell/myeloma fusions with granulocyte macrophage colony-stimulating factor (GM-CSF) adjuvant plus lenalidomide maintenance therapy versus maintenance therapy alone or with GM-CSF following autologous transplant as part of upfront treatment of multiple myeloma (MM). It is hypothesized that the dendritic cell myeloma vaccine will result in improved response in patients with multiple myeloma after autologous Hematopoietic Cell Transplant (HCT).

DETAILED DESCRIPTION:
The study is a three-arm, phase II randomized, open-labeled clinical trial that randomizes patients to vaccination with Dendritic Cell (DC)/myeloma fusions/GM-CSF plus lenalidomide maintenance therapy or lenalidomide maintenance therapy with or without GM-CSF following autologous transplant as part of upfront treatment for patients diagnosed with multiple myeloma. Patients are randomized approximately 2 months post transplant and will begin maintenance lenalidomide between day 90 and 100. The primary objective of this randomized trial is to compare the proportion of patients alive and in complete response (defined as CR or sCR) at one year post transplant between patients receiving DC/myeloma vaccine/GM-CSF with lenalidomide maintenance therapy to those receiving lenalidomide maintenance therapy with or without GM-CSF.

ELIGIBILITY:
Initial Inclusion Criteria:

1. Patients must be considered transplant eligible by the treating physician at time of study entry.
2. Patients must meet the criteria for symptomatic multiple myeloma prior to initiating systemic anti-myeloma treatment.
3. Age >18 years and ≤ 70 years at the time of enrollment
4. Karnofsky Performance status of ≥ 70%
5. Patients must have > 20% plasma cells in the bone marrow aspirate differential <60 days prior to enrollment. The required bone marrow evaluation will need to be repeated for patients who received more than 1 cycle of anti-myeloma therapy (corticosteroid with or without other anti-myeloma agents)
6. Patients must have received ≤ 1 cycles of systemic anti-myeloma therapy.
7. Renal: Creatinine clearance of ≥ 40 mL/min, estimated or calculated.

Initial Exclusion Criteria:

1. Patients with a prior autologous or allogeneic HCT
2. Patients with purely non-secretory MM [absence of a monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques and the absence of involved serum free light chain >100 mg/L]. Patients with light chain MM detected in the serum by free light chain assay are eligible.
3. Patients with Plasma Cell Leukemia
4. Patients with disease progression prior to enrollment
5. Patients seropositive for the human immunodeficiency virus (HIV).
6. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening will be documented by the investigator as not medically relevant.
7. Patients with active clinically significant autoimmune disease, defined as a history of requiring systemic immunosuppressive therapy and at ongoing risk for potential disease exacerbation. Patients with a history of autoimmune thyroid disease, asthma, or limited skin manifestations are potentially eligible.
8. Patients receiving other investigational immunotherapy or anti-myeloma drugs within 14 days before enrollment.
9. Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent < 5 years prior to enrollment will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs. Cancer treated with curative intent > 5 years prior to enrollment is allowed.
10. Female patients who are pregnant (positive beta-HCG) or breastfeeding.
11. Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use contraceptive techniques (Appendix D) during the length of lenalidomide maintenance therapy.
12. Patients who have received mid-intensity melphalan (>50 mg IV) as part of prior therapy.
13. Prior organ transplant requiring immunosuppressive therapy.
14. Patients who previously received lenalidomide and have experienced toxicities resulting in treatment discontinuation.
15. Patients who experienced thromboembolic events while on full anticoagulation during prior therapy with lenalidomide or thalidomide.
16. Patients unwilling to take deep vein thrombosis (DVT) prophylaxis.
17. Patients unable or unwilling to provide informed consent.
18. Patients unable or unwilling to return to the transplant center for their assigned treatments.

Randomization Inclusion Criteria:

1. Patient received transplant < 12 months of enrollment onto BMT CTN 1401.
2. No disease progression since initiation of systemic anti-myeloma therapy as determined within seven days of randomization/enrollment.
3. Received an autologous cell transplant with melphalan 200mg/m^2 with a minimum cell dose of 2x10^6 CD34+ cells/kg (actual body weight).
4. Mucositis and gastrointestinal symptoms resolved, off hyperalimentation and intravenous hydration.
5. No evidence of uncontrolled infection requiring systemic therapy. Patients who completed treatment for an infection but are continuing antibiotics, anti-viral, or anti-fungal therapy for prophylaxis are eligible to continue on protocol.
6. Platelet count ≥75,000/mm^3 (without transfusion in previous 7 days).
7. Absolute neutrophil count (ANC) ≥ 1,500/mm^3 without filgrastim administration within 7 days, or pegfilgrastim within 14 days of measurement.
8. Hepatic: bilirubin < 2x the upper limit of normal and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5x the upper limit of normal. (Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value of 2x the upper limit of normal)
9. Renal: Creatinine clearance of ≥ 40 mL/min, estimated or calculated. Patients with creatinine clearance ≥30 but <40 will be considered with review/approval from the protocol chairs or officer if the cause of renal insufficiency is associated with multiple myeloma.
10. All study participants must be registered into the mandatory Revlimid REMs program, and be willing and able to comply with the requirements.
11. Females of childbearing potential (FCBP) as defined in section 2.7.1.1 must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days)
12. FCBP must either commit to abstain continuously from sexual intercourse or use TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide, during therapy, during dose interruptions, and continuing for 4 weeks following discontinuation of lenalidomide.
13. FCBP must agree to ongoing pregnancy testing as required by the Revlimid REMs program.
14. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy while taking lenalidomide, during dose interruptions and for 28 days after discontinuing lenalidomide.
15. Patients must be willing to receive DVT prophylaxis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (15):
- United States (15):
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center/Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State University/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Chung DJ, Shah N, Wu J, Logan B, Bisharat L, Callander N, Cheloni G, Anderson K, Chodon T, Dhakal B, Devine S, Somaiya Dutt P, Efebera Y, Geller N, Ghiasuddin H, Hematti P, Holmberg L, Howard A, Johnson B, Karagkouni D, Lazarus HM, Malek E, McCarthy P, McKenna D, Mendizabal A, Nooka A, Munshi N, O'Donnell L, Rapoport AP, Reese J, Rosenblatt J, Soiffer R, Stroopinsky D, Uhl L, Vlachos IS, Waller EK, Young JW, Pasquini MC, Avigan D. Randomized Phase II Trial of Dendritic Cell/Myeloma Fusion Vaccine with Lenalidomide Maintenance after Upfront Autologous Hematopoietic Cell Transplantation for Multiple Myeloma: BMT CTN 1401. Clin Cancer Res. 2023 Dec 1;29(23):4784-4796. doi: 10.1158/1078-0432.CCR-23-0235. PMID 37463058
- See also: Blood and Marrow Transplant Clinical Trials Network — http://bmtctn.net/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on July 25, 2016 and closed to accrual on October 12, 2018 with 203 participants enrolled from 18 participating centers. The final study database lock was done September 9, 2021.
Pre-assignment Details: Sixty-three participants dropped out of the study prior to randomization and 140 participants received a transplant and proceeded to randomization. The reasons for dropout include insufficient tumor cells collected (n=13), withdrew consent from study (n=12), ineligible to be randomized (n=8), disease progression prior to randomization (n=6), refused or did not make it to transplantation (n=10), physician decision (n=7), manufacturing failure (n=4), lost to follow up (n=2), and insurance (n=1).
Groups:
- Lenalidomide, Vaccine, and GM-CSF: Patients will undergo tumor cell collection and autologous stem cell transplant with melphalan. Patients will undergo leukapheresis and then will receive maintenance lenalidomide with myeloma vaccine and GM-CSF.
  Tumor Cell Collection: Patients will undergo aspiration of 30 mL of bone marrow from which myeloma cell will be isolated and frozen for subsequent vaccine generation.
  Autologous Stem Cell Transplant: Patients will receive an autologous graft of a minimum cell dose of 2.0 x 10^6 CD34+ cells/kg patient actual body weight per transplantation with high-dose melphalan of 200mg/m^2 at the schedule and timing according to institutional practices.
  Leukapheresis: Blood samples will be collected through a catheter in the neck or chest and leukapheresis will be performed using standard clinical procedures.
  Lenalidomide: Maintenance therapy with lenalidomide will begin between 90 and 100 days after stem cell infusion. Lenalidomide will be administered initially at a dose of 10 mg per day continuously. Cycle duration during maintenance therapy is 28 days. Patients will continue lenalidomide for two years from initiation of therapy.
  Myeloma vaccine: The target dose is 3 x 10^6 fusion cells per vaccine. A minimum of 3 x 10^6 total fusion cells will be required to proceed with vaccine administration. Patients will receive the DC/MM fusion vaccine on day 1 of cycles 2, 3, and 4 of lenalidomide maintenance.
  GM-CSF: 100 ug GM-CSF will be given for a total of 4 days of each cycle.
Period: Overall Study
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Started | 68 | 37 | 35
Completed | 61 | 33 | 30
Not Completed | 7 | 4 | 5
Not completed — Death | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 3
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Investigational study drug permanently discontinued | 3 | 1 | 0
Not completed — Covid | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide | Total
Number analyzed (Participants) | 68 | 37 | 35 | 140
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [41.6 to 70.2] | 62.3 [44.2 to 70.2] | 59.1 [35.2 to 70.9] | 60.0 [35.2 to 70.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 18 | 63
  Male | 41 | 19 | 17 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 11
  Not Hispanic or Latino | 61 | 33 | 30 | 124
  Unknown or Not Reported | 3 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 5 | 15
  White | 54 | 30 | 28 | 112
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 2 | 8
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    100 | 16 | 7 | 9 | 32
    90 | 29 | 10 | 14 | 53
    80 | 17 | 15 | 9 | 41
    70 | 6 | 5 | 3 | 14
Disease Response at Randomization [Count of Participants; unit: Participants] — CR: no original monoclonal paraprotein, < 5% BM plasma cells, no lytic bone lesions increase, and no soft tissue plasmacytomas. sCR: CR, normal FLC ratio, and no clonal cells. PR: >= 50% serum monoclonal paraprotein decrease and 24 hr urinary monoclonal decrease, or >= 50% involved and uninvolved FLC decrease or a 50% decrease in involved FLC w/ 50% ratio decrease, or >= 50% BM plasma cells decrease, or >= 50% soft tissue plasmacytomas decrease. VGPR: PR, paraprotein decrease or >= 90% serum paraprotein decrease, and a 90% involved light chain decrease. SD: none of above and no progression.
  Participants
    Stringent Complete Response (sCR) | 11 | 6 | 4 | 21
    Complete Response (CR) | 11 | 9 | 9 | 29
    Very Good Partial Response (VGPR) | 37 | 15 | 17 | 69
    Partial Response (PR) | 9 | 7 | 5 | 21
    Stable Response | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 1-year Response Rate of CR/sCR
Description: The primary objective of this randomized trial is to compare the proportion of patients alive and in complete response (CR or sCR) at one year post transplant between patients receiving DC/myeloma vaccine/GM-CSF with lenalidomide maintenance therapy to those receiving lenalidomide maintenance therapy with or without GM-CSF. Complete Response (CR) is defined to require all the followings: Absence of the original monoclonal paraprotein in serum and urine by routine electrophoresis and by immunofixation; Less than 5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy, if biopsy is performed; No increase in size or number of lytic bone lesions on radiological investigations; Disappearance of soft tissue plasmacytomas. Stringent Complete Response (sCR) is defined to require all the followings in addition to CR: Normal free light chain ratio (FLC); Absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Time Frame: 1 year
Population: The primary analysis population includes all the randomized participants. Protocol defines primary analysis is to compare participants receiving vaccine vs those without vaccine. So no vaccine arms with or without GM-CSF are combined. Four participants withdrew consent to all study procedures before 1-year post-transplant. Of these, 2 cases on the Lenalidomide/GM-CSF arm and 2 cases on the Lenalidomide Alone arm. These participants were not evaluable for the primary endpoint and ERC confirmed.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Lenalidomide With or Without GM-CSF: Patients will undergo tumor cell collection and autologous stem cell transplant with melphalan. Patients will receive maintenance lenalidomide with or without GM-CSF.
  Tumor Cell Collection: Patients will undergo aspiration of 30 mL of bone marrow from which myeloma cell preparations will be generated. Myeloma cells will be isolated and frozen for subsequent vaccine generation for patients randomized to the vaccine arm (randomization occurs after transplant and recovery).
  Autologous Stem Cell Transplant: Patients will receive an autologous graft with a minimum cell dose of 2.0 x 10^6 CD34+ cells/kg patient actual body weight per autologous transplantation.
  Melphalan: Autologous hematopoietic cell transplant will be done with high-dose melphalan of 200mg/m^2 at the schedule and timing according to institutional practices.
  Lenalidomide: Maintenance therapy with lenalidomide will begin between 90 and 100 days after stem cell infusion. Lenalidomide will be administered initially at a dose of 10 mg per day continuously. Cycle duration during maintenance therapy is 28 days. Patients will continue lenalidomide for two years from initiation of therapy.
  GM-CSF: 100 ug GM-CSF will be given subcutaneously in the upper thigh and daily for a total of 4 days of each cycle.
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 68
percentage of participants | 52.9 [44.5 to 61.3] | 50.0 [41.6 to 58.4]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The proportion of patients alive and in CR/sCR at 1 year post transplant will be described in the vaccine and no vaccine groups with 80% confidence intervals and compared between groups using a two-sample Z test comparing binomial proportions; Test type: Superiority; p = 0.3657, Z test — A one-sided significance level of 0.10 is used to assess whether the vaccine appears promising relative to control; difference in the proportions = 2.9, 80% CI 2-sided [-8.8 to 14.6]
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; A secondary analysis stratified on disease response prior to randomization between arms will be conducted using a Cochran-Mantel-Haenszel test, and a stratified odds ratio along with 80% confidence intervals will be estimated; Test type: Equivalence — The stratified odds ratio is estimated with 80% confidence intervals; p = 0.7461, Cochran-Mantel-Haenszel — P-value is provided by Breslow-Day Test for Homogeneity of the Odds Ratios; Odds Ratio (OR) = 1.19, 80% CI 2-sided [0.70 to 2.03] — The Cochran-Mantel-Haenszel Odds Ratio estimate is for the Stratification. Stratum 1 is sCR/CR at Randomization. Stratum 2 is VGPR/PR/Stable Response at Randomization
Statistical Analysis 3: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; A secondary pairwise analysis of CR/sCR rates comparing the vaccine arm to Lenalidomide/GM-CSF arm at 1 year post transplant; Test type: Superiority — The proportion of patients alive and in CR/sCR at 1 year post transplant will be compared in the vaccine arm to Lenalidomide/GM-CSF arm with 80% confidence intervals using a two-sample Z test comparing binomial proportions; p = 0.2429, Z test; difference in the proportions = 7.2, 80% CI 2-sided [-6.4 to 20.6]
Statistical Analysis 4: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; A secondary pairwise analysis of CR rates comparing the vaccine arm to Lenalidomide alone arm at 1 year post transplant; Test type: Superiority — The proportion of patients alive and in CR/sCR at 1 year post transplant will be compared in the vaccine arm to Lenalidomide alone arm with 80% confidence intervals using a two-sample Z test comparing binomial proportions; p = 0.4397, Z test; difference in the proportions = -1.6, 80% CI 2-sided [-15.6 to 12.4]

2. Secondary Outcome: Participants Response to Treatment
Description: A participant's disease status is evaluated based on the International Uniform Response Criteria per protocol. Before disease progression (PD), all disease classifications including stringent complete response (sCR), complete response (CR), very good partial remission (VGPR), partial response (PR), stable disease (SD) are relative to participant's disease status at study entry. Disease status is 'Not Evaluable' when disease assessment is not required, or disease status is missing.
Time Frame: 6 months, 1 year, and 2 years post-transplant and at Cycles 3(Day 57), 6(Day 141), 9(Day 225), 12(Day 309), 15 (Day 393), 18(Day 477), 21(Day 561) and 24(Day 654) of maintenance therapy
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
Participants
  Disease Status at 6 Months: Stringent Complete Response (sCR) | 12 | 9 | 8
  Disease Status at 6 Months: Complete Response (CR) | 17 | 8 | 10
  Disease Status at 6 Months: Very Good Partial Remission (VGPR) | 28 | 12 | 13
  Disease Status at 6 Months: Partial Response (PR) | 5 | 5 | 2
  Disease Status at 6 Months: Stable Disease (SD) | 2 | 1 | 0
  Disease Status at 6 Months: Progression (PD) | 0 | 0 | 0
  Disease Status at 6 Months: Dead | 0 | 0 | 0
  Disease Status at 6 Months: Not Evaluable | 4 | 2 | 2
  Disease Status at 12 Months: Stringent Complete Response (sCR) | 18 | 8 | 9
  Disease Status at 12 Months: Complete Response (CR) | 18 | 8 | 9
  Disease Status at 12 Months: Very Good Partial Remission (VGPR) | 22 | 12 | 10
  Disease Status at 12 Months: Partial Response (PR) | 4 | 7 | 3
  Disease Status at 12 Months: Stable Disease (SD) | 0 | 0 | 0
  Disease Status at 12 Months: Progression (PD) | 5 | 0 | 2
  Disease Status at 12 Months: Dead | 1 | 0 | 0
  Disease Status at 12 Months: Not Evaluable | 0 | 2 | 2
  Disease Status at 24 Months: Stringent Complete Response (sCR) | 17 | 7 | 9
  Disease Status at 24 Months: Complete Response (CR) | 13 | 6 | 10
  Disease Status at 24 Months: Very Good Partial Remission (VGPR) | 15 | 15 | 3
  Disease Status at 24 Months: Partial Response (PR) | 6 | 4 | 2
  Disease Status at 24 Months: Stable Disease (SD) | 0 | 0 | 0
  Disease Status at 24 Months: Progression (PD) | 2 | 0 | 0
  Disease Status at 24 Months: Dead | 2 | 0 | 1
  Disease Status at 24 Months: Not Evaluable | 13 | 5 | 10
  Disease Status at Cycle 3 (Day 57 Assessment): Stringent Complete Response (sCR) | 8 | 9 | 7
  Disease Status at Cycle 3 (Day 57 Assessment): Complete Response (CR) | 19 | 5 | 14
  Disease Status at Cycle 3 (Day 57 Assessment): Very Good Partial Remission (VGPR) | 35 | 15 | 11
  Disease Status at Cycle 3 (Day 57 Assessment): Partial Response (PR) | 5 | 6 | 2
  Disease Status at Cycle 3 (Day 57 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 3 (Day 57 Assessment): Progression (PD) | 0 | 0 | 0
  Disease Status at Cycle 3 (Day 57 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 3 (Day 57 Assessment): Not Evaluable | 1 | 2 | 1
  Disease Status at Cycle 6 (Day 141 Assessment): Stringent Complete Response (sCR) | 13 | 7 | 7
  Disease Status at Cycle 6 (Day 141 Assessment): Complete Response (CR) | 18 | 7 | 14
  Disease Status at Cycle 6 (Day 141 Assessment): Very Good Partial Remission (VGPR) | 28 | 14 | 10
  Disease Status at Cycle 6 (Day 141 Assessment): Partial Response (PR) | 6 | 7 | 2
  Disease Status at Cycle 6 (Day 141 Assessment): Stable Disease (SD) | 1 | 0 | 0
  Disease Status at Cycle 6 (Day 141 Assessment): Progression (PD) | 1 | 0 | 0
  Disease Status at Cycle 6 (Day 141 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 6 (Day 141 Assessment): Not Evaluable | 1 | 2 | 2
  Disease Status at Cycle 9 (Day 225 Assessment): Stringent Complete Response (sCR) | 16 | 8 | 9
  Disease Status at Cycle 9 (Day 225 Assessment): Complete Response (CR) | 17 | 7 | 15
  Disease Status at Cycle 9 (Day 225 Assessment): Very Good Partial Remission (VGPR) | 24 | 13 | 7
  Disease Status at Cycle 9 (Day 225 Assessment): Partial Response (PR) | 6 | 7 | 2
  Disease Status at Cycle 9 (Day 225 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 9 (Day 225 Assessment): Progression (PD) | 2 | 0 | 0
  Disease Status at Cycle 9 (Day 225 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 9 (Day 225 Assessment): Not Evaluable | 3 | 2 | 2
  Disease Status at Cycle 12 (Day 309 Assessment): Stringent Complete Response (sCR) | 18 | 9 | 9
  Disease Status at Cycle 12 (Day 309 Assessment): Complete Response (CR) | 18 | 6 | 10
  Disease Status at Cycle 12 (Day 309 Assessment): Very Good Partial Remission (VGPR) | 20 | 13 | 7
  Disease Status at Cycle 12 (Day 309 Assessment): Partial Response (PR) | 5 | 7 | 4
  Disease Status at Cycle 12 (Day 309 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 12 (Day 309 Assessment): Progression (PD) | 0 | 0 | 2
  Disease Status at Cycle 12 (Day 309 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 12 (Day 309 Assessment): Not Evaluable | 7 | 2 | 3
  Disease Status at Cycle 15 (Day 393 Assessment): Stringent Complete Response (sCR) | 18 | 9 | 9
  Disease Status at Cycle 15 (Day 393 Assessment): Complete Response (CR) | 17 | 5 | 13
  Disease Status at Cycle 15 (Day 393 Assessment): Very Good Partial Remission (VGPR) | 18 | 11 | 6
  Disease Status at Cycle 15 (Day 393 Assessment): Partial Response (PR) | 4 | 7 | 2
  Disease Status at Cycle 15 (Day 393 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 15 (Day 393 Assessment): Progression (PD) | 3 | 0 | 1
  Disease Status at Cycle 15 (Day 393 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 15 (Day 393 Assessment): Not Evaluable | 8 | 5 | 4
  Disease Status at Cycle 18 (Day 477 Assessment): Stringent Complete Response (sCR) | 20 | 7 | 7
  Disease Status at Cycle 18 (Day 477 Assessment): Complete Response (CR) | 16 | 7 | 13
  Disease Status at Cycle 18 (Day 477 Assessment): Very Good Partial Remission (VGPR) | 17 | 14 | 6
  Disease Status at Cycle 18 (Day 477 Assessment): Partial Response (PR) | 3 | 6 | 1
  Disease Status at Cycle 18 (Day 477 Assessment): Stable Disease (SD) | 2 | 0 | 0
  Disease Status at Cycle 18 (Day 477 Assessment): Progression (PD) | 1 | 0 | 1
  Disease Status at Cycle 18 (Day 477 Assessment): Dead | 0 | 0 | 0
  Disease Status at Cycle 18 (Day 477 Assessment): Not Evaluable | 9 | 3 | 7
  Disease Status at Cycle 21 (Day 561 Assessment): Stringent Complete Response (sCR) | 20 | 6 | 10
  Disease Status at Cycle 21 (Day 561 Assessment): Complete Response (CR) | 15 | 5 | 11
  Disease Status at Cycle 21 (Day 561 Assessment): Very Good Partial Remission (VGPR) | 14 | 17 | 6
  Disease Status at Cycle 21 (Day 561 Assessment): Partial Response (PR) | 5 | 4 | 1
  Disease Status at Cycle 21 (Day 561 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 21 (Day 561 Assessment): Progression (PD) | 2 | 0 | 0
  Disease Status at Cycle 21 (Day 561 Assessment): Dead | 1 | 0 | 0
  Disease Status at Cycle 21 (Day 561 Assessment): Not Evaluable | 11 | 5 | 7
  Disease Status at Cycle 24 (Day 654 Assessment): Stringent Complete Response (sCR) | 19 | 6 | 9
  Disease Status at Cycle 24 (Day 654 Assessment): Complete Response (CR) | 15 | 7 | 11
  Disease Status at Cycle 24 (Day 654 Assessment): Very Good Partial Remission (VGPR) | 14 | 16 | 6
  Disease Status at Cycle 24 (Day 654 Assessment): Partial Response (PR) | 6 | 3 | 1
  Disease Status at Cycle 24 (Day 654 Assessment): Stable Disease (SD) | 0 | 0 | 0
  Disease Status at Cycle 24 (Day 654 Assessment): Progression (PD) | 1 | 1 | 0
  Disease Status at Cycle 24 (Day 654 Assessment): Dead | 1 | 0 | 1
  Disease Status at Cycle 24 (Day 654 Assessment): Not Evaluable | 12 | 4 | 7
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine and the combined non-vaccine arms at 6 months Post Transplant; Test type: Superiority; p = 0.9376, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide/GM-CSF arm at 6 months Post Transplant; Test type: Superiority; p = 0.4887, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide alone arm at 6 months Post Transplant; Test type: Superiority; p = 0.5176, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 4: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between lenalidomide/GM-CSF arm and lenalidomide alone arm at 6 months Post Transplant; Test type: Superiority; p = 0.2461, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 5: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine and the combined non-vaccine arms at 1 year Post Transplant; Test type: Superiority; p = 0.2530, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 6: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide/GM-CSF arm at 1 year Post Transplant; Test type: Superiority; p = 0.2213, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 7: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide alone arm at 1 year Post Transplant; Test type: Superiority; p = 0.4930, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 8: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the lenalidomide/GM-CSF arm and lenalidomide alone arm at 1 year Post Transplant; Test type: Superiority; p = 0.6591, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 9: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine and the combined non-vaccine arms at 2 years Post Transplant; Test type: Superiority; p = 0.6790, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 10: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide/GM-CSF arm at 2 years Post Transplant; Test type: Superiority; p = 0.3124, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 11: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the vaccine arm and lenalidomide alone arm at 2 years Post Transplant; Test type: Superiority; p = 0.7379, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 12: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; In this pairwise analysis, the proportion of participants alive and with sCR/CR/VGPR will be compared between the lenalidomide/GM-CSF arm and lenalidomide alone arm at 2 years Post Transplant; Test type: Superiority; p = 0.2379, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 13: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; Proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between the vaccine and the combined non-vaccine arms at 6 months Post Transplant; Test type: Superiority; p = 0.5353, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 14: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; Proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between the vaccine and the combined non-vaccine arms at 12 months Post Transplant; Test type: Superiority; p = 0.4417, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 15: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF vs Maintenance Lenalidomide; Proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between the vaccine and the combined non-vaccine arms at 24 months Post Transplant; Test type: Superiority; p = 0.9450, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 16: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; A pairwise analysis of proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between the vaccine arm and lenalidomide/GM-CSF arm is conducted at 1 year post transplant; Test type: Superiority; p = 0.1599, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 17: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; A pairwise analysis of proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between the vaccine arm and lenalidomide alone arm is conducted at 1 year post transplant; Test type: Superiority; p = 0.8984, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 18: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; A pairwise analysis of proportion of participants achieving CR among the subset of participants who are not in CR at the time of randomization between lenalidomide/GM-CSF arm and lenalidomide alone arm is conducted at 1 year post transplant; Test type: Superiority; p = 0.1757, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05

3. Secondary Outcome: Percentage of Participants With Myeloma Progression of Vaccine and Non-vaccine Arms
Description: The event for this endpoint is defined as disease progression from CR/sCR or progressive disease for participants not in CR/sCR, or initiation of off protocol antimyeloma therapy. The cumulative incidence of myeloma progression will be compared between the vaccine arm and the combined non-vaccine arms using Gray's test and treating death (without documentation of disease progression) as a competing risk. Participants alive without disease progression at last observation will be censored at the date of last contact.
Time Frame: 2 years
Population: The randomized participants are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
percentage of participants | 20.7 [12 to 31.1] | 11.8 [5.5 to 20.7]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of Myeloma Progression between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.161, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

4. Secondary Outcome: Percentage of Participants With Myeloma Progression in Pairwise Analysis
Description: This is the pairwise comparison for percentage of participants with Myeloma Progression. The event for this endpoint is defined as disease progression from CR/sCR or progressive disease for participants not in CR/sCR, or initiation of off protocol antimyeloma therapy. The cumulative incidence of myeloma progression will be compared between the vaccine arm, lenalidomide/GM-CSF arm and lenalidomide alone arm using Gray's test and treating death (without documentation of disease progression) as a competing risk. Participants alive without disease progression at last observation will be censored at the date of last contact.
Time Frame: 2 years
Population: The randomized participants are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
percentage of participants | 20.7 [12 to 31.1] | 8.7 [2.2 to 21.0] | 15.1 [5.4 to 29.4]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; The null hypothesis is that there is no difference of Myeloma Progression between the vaccine arm and lenalidomide/GM-CSF arm; Test type: Superiority; p = 0.116, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Myeloma Progression between the vaccine arm and lenalidomide alone arm; Test type: Superiority; p = 0.519, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Myeloma Progression between the lenalidomide/GM-CSF arm and lenalidomide alone arm; Test type: Superiority; p = 0.387, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

5. Secondary Outcome: Percentage of Participants With Treatment-related Mortality (TRM)
Description: TRM is defined as death occurring in a patient from causes other than disease relapse or progression. Disease progression is the competing event for TRM. Patients alive without disease progression at last contact are considered censored for this event. TRM from time of randomization will be compared between vaccine and no-vaccine arms combined starting at time of randomization.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
percentage of participants | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Percentage of Participants With Progression-Free Survival
Description: Death or disease progression will be considered as events for this endpoint. The time to event will be calculated as time from randomization to disease progression, death, initiation of non-protocol anti-myeloma therapy, loss to follow-up or the end of the study, whichever comes first. The Kaplan-Meier estimator will be constructed for each treatment arm. Progression-free survival was compared between the vaccine and the combined non-vaccine arms using the log-rank test.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
percentage of participants | 79.3 [67.6 to 87.2] | 88.2 [77.8 to 93.3]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of Progression-Free Survival between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.168, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

7. Secondary Outcome: Percentage of Participants With Progression-Free Survival in Pairwise Analysis
Description: This is the pairwise comparison for percentage of participants with Progression-Free Survival. Death or disease progression will be considered as events for this endpoint. The time to event will be calculated as time from randomization to disease progression, death, initiation of non-protocol anti-myeloma therapy, loss to follow-up or the end of the study, whichever comes first. The Kaplan-Meier estimator will be constructed for each treatment arm. Progression-free survival was compared between the vaccine arm, lenalidomide/GM-CSF arm and lenalidomide alone arm.
Time Frame: 2 year
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
percentage of participants | 79.3 [67.6 to 87.2] | 91.3 [75.5 to 97.1] | 84.9 [67.5 to 93.4]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; The null hypothesis is that there is no difference of Progression-Free Survival between the vaccine arm and lenalidomide/GM-CSF arm; Test type: Superiority; p = 0.120, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Progression-Free Survival between the vaccine arm and lenalidomide alone arm; Test type: Superiority; p = 0.519, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Progression-Free Survival between the lenalidomide/GM-CSF arm and lenalidomide alone arm; Test type: Superiority; p = 0.387, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

8. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Death from any cause is considered as events for this endpoint. The time to event is calculated as time from randomization to death, loss to follow-up or the end of the study, whichever comes first. Patients alive at the time of last observation are considered censored. The Kaplan-Meier estimator will be constructed for each treatment arm. Overall survival are compared between the vaccine and the combined non-vaccine arms from time of randomization.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
percentage of participants | 97 [88.6 to 99.2] | 98.5 [89.7 to 99.8]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of overall Survival between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.563, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

9. Secondary Outcome: Percentage of Participants With Overall Survival in Pairwise Analysis
Description: This is the pairwise comparison for percentage of participants with Overall Survival. Death from any cause is considered as events for this endpoint. The time to event is calculated as time from randomization to death, loss to follow-up or the end of the study, whichever comes first. Patients alive at the time of last observation are considered censored. The Kaplan-Meier estimator will be constructed for each treatment arm. Overall survival are compared between the vaccine arm, lenalidomide/GM-CSF arm and lenalidomide alone arm from time of randomization.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
percentage of participants | 97 [88.6 to 99.2] | 100 [100 to 100] | 96.9 [79.8 to 99.6]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; The null hypothesis is that there is no difference of overall Survival between the vaccine arm and lenalidomide/GM-CSF arm; Test type: Superiority; p = 0.308, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of overall Survival between the vaccine arm and lenalidomide alone arm; Test type: Superiority; p = 0.990, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of overall Survival between the lenalidomide/GM-CSF arm and lenalidomide alone arm; Test type: Superiority; p = 0.303, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

10. Secondary Outcome: Number of Grade ≥ 3 Toxicities
Description: Toxicities are evaluated using NCI CTCAE version 4.0 at pre-maintenance initiation and during maintenance therapy monthly for the first 4 cycles and then at cycles 6, 9, 15, 21, 24, which correspond to Day 1, 29, 57, 85, 141, 225, 393, 561, and 645 post maintenance initiation. All Grade ≥ 3 toxicities will be tabulated for treatment arms. Toxicities are categorized by organ system according to the CTCAE. Toxicities that involve multiple questions per organ system are combined in one category.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number; unit: Toxicities
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
Toxicities
  Auditory Disorders | 1 | 0 | 0
  Blood and Lymphatic Disorders | 81 | 40 | 38
  Cardiovascular Disorders | 4 | 3 | 2
  GI Disorders | 15 | 4 | 2
  General Disorders | 5 | 2 | 2
  Hepatobiliary/Pancreas Disorders | 4 | 1 | 1
  Immune System Disorders | 2 | 0 | 0
  Investigations | 2 | 0 | 1
  Metabolism and Nutrition Disorders | 7 | 1 | 3
  Musculoskeletal and Connective Tissue Disorders | 1 | 1 | 2
  Nervous System Disorders | 14 | 5 | 1
  Renal Disorders | 1 | 0 | 2
  Respiratory, Thoracic and Mediastinal Disorders | 5 | 1 | 2
  Skin and Subcutaneous Tissue Disorders | 4 | 5 | 7
  Vascular Disorders | 6 | 11 | 3
  Abnormal Liver Symptoms | 0 | 1 | 0

11. Secondary Outcome: Participants With Grade ≥ 3 Toxicities
Description: Toxicities are evaluated using NCI CTCAE version 4.0 at pre-maintenance initiation and during maintenance therapy monthly for the first 4 cycles and then at cycles 6, 9, 15, 21, 24, which correspond to Day 1, 29, 57, 85, 141, 225, 393, 561, and 645 post maintenance initiation. The number of participants experiencing Grade ≥ 3 toxicity are displayed for the vaccine and non-vaccine arms separately. The proportion of participants experiencing Grade ≥ 3 toxicity are compared between the vaccine and non-vaccine arms combined.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
Participants | 53 | 49
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of proportions of patients With Grade ≥ 3 Toxicities between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.189, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05

12. Secondary Outcome: Number of Grade 2 and 3 Infections
Description: Grade 2 and 3 infections, as defined by the BMT CTN Technical MOP, occurring after randomization will be reported. The incidence of definite and probable viral, fungal and bacterial infections will be tabulated for each patient.
Time Frame: 2years
Population: The randomized participants are included in the analysis
Measure: Number; unit: infections
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
infections
  Bacterial | 10 | 3 | 6
  Viral | 14 | 6 | 14
  Fungal | 0 | 0 | 0
  Other | 1 | 0 | 1

13. Secondary Outcome: Percentage of Participants With Grade 2 and 3 Infections
Description: Grade 2 and 3 infections, as defined by the BMT CTN Technical MOP, are reported on the study. The cumulative incidence of infections post randomization, treating death as a competing risk, were compared between the vaccine and the combined non-vaccine groups using the Gray's test.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 68 | 72
percentage of participants | 26.6 [16.7 to 37.6] | 23.2 [14 to 33.8]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of Participants with Grade 2 and 3 infections between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.82, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

14. Secondary Outcome: Percentage of Participants With Grade 2 and 3 Infections in Pairwise Analysis
Description: This is the pairwise comparison for percentage of participants with Grade 2 and 3 infections. Grade 2 and 3 infections, as defined by the BMT CTN Technical MOP, are reported on the study. The cumulative incidence of infections post randomization, treating death as a competing risk, were compared between the vaccine arm, lenalidomide/GM-CSF arm and lenalidomide alone arm using the Gray's test.
Time Frame: 2 years
Population: The randomized participants are included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
Number analyzed (Participants) | 68 | 37 | 35
percentage of participants | 26.6 [16.7 to 37.6] | 14.2 [5.1 to 27.8] | 32.6 [17.5 to 48.7]
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide and GM-CSF; The null hypothesis is that there is no difference of Participants with Grade 2 and 3 infections between the vaccine arm and lenalidomide/GM-CSF arm; Test type: Superiority; p = 0.21, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Participants with Grade 2 and 3 infections between the vaccine arm and lenalidomide alone arm; Test type: Superiority; p = 0.40, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Lenalidomide and GM-CSF vs Maintenance Lenalidomide; The null hypothesis is that there is no difference of Participants with Grade 2 and 3 infections between the lenalidomide/GM-CSF arm and lenalidomide alone arm; Test type: Superiority; p = 0.08, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

15. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD)
Description: Minimal residual disease (MRD) is defined as the presence of malignant plasma cells detected by multicolor flow cytometry among patients who are in complete remission. Multichannel flow cytometry will be used to establish MRD based on the presence of malignant plasma cells that are CD45 (-/dim), CD38+, CD138+, CD19-, CD56+ kappa or lambda restricted. The number of patients with MRD negative (MRD-) are described using frequencies at pre-randomization and 9th cycle post-randomization and compared between the vaccine arm with the no-vaccine arms combined.
Time Frame: Pre-randomization, Post-randomization at Cycle 9
Population: The randomized participants who had MRD assessment. Participants who did not have MRD assessment are not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide With or Without GM-CSF
Number analyzed (Participants) | 65 | 66
Participants
  Pre-randomization | 35 | 31
  Post-randomization at Cycle 9: number analyzed (Participants) | 53 | 59
  Post-randomization at Cycle 9 | 38 | 41
Statistical Analysis 1: Comparison: Lenalidomide, Vaccine, and GM-CSF vs Lenalidomide With or Without GM-CSF; The null hypothesis is that there is no difference of proportions of patients without Minimal Residual Disease between vaccine vs. non- vaccine arms; Test type: Superiority; p = 0.80, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lenalidomide, Vaccine, and GM-CSF | Lenalidomide and GM-CSF | Maintenance Lenalidomide
All-Cause Mortality (participants affected / at risk) | 3/68 | 0/37 | 1/35
Serious Adverse Events (participants affected / at risk) | 2/68 | 3/37 | 1/35
Other Adverse Events (participants affected / at risk) | 3/68 | 3/37 | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide, Vaccine, and GM-CSF (N=68) | Lenalidomide and GM-CSF (N=37) | Maintenance Lenalidomide (N=35)
NEUTROPENIC FEVER (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PROLONGED QTC (Investigations) | 1 (1) | 0 (0) | 0 (0)
ELEVATE LIVER ENZYMES (Investigations) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TESTS INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide, Vaccine, and GM-CSF (N=68) | Lenalidomide and GM-CSF (N=37) | Maintenance Lenalidomide (N=35)
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ELEVATED ALT (Investigations) | 1 (1) | 0 (0) | 0 (0)
INCREASED ALT > 3.0 X ULN (Investigations) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ELEVATED LFT (Investigations) | 0 (0) | 0 (0) | 1 (1)
GRADE 2 DVT (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
GRADE 2 TRANSAMINITIS (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT02728102/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT02728102/SAP_003.pdf
  • Informed Consent Form (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT02728102/ICF_002.pdf